CLINICAL TRIAL: NCT03101020
Title: Visceral Manipulation in Patients With Chronic Low Back Pain: Randomized Controlled Trial
Brief Title: Visceral Manipulation in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sorocaba (Other)
Responsible Party: Principal Investigator, Luciane Cruz Lopes, Director, Clinical Research, University of Sorocaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Visceral Mob and LBP
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Chronic Low Back Pain
Keywords: Visceral Manipulation

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will receive standard care physiotherapy for low back pain according to the evidence presented in the study of Delitto et al. The care includes advice for correct postures to perform daily activities; abdominal, pelvic and lumbar muscles re-training and strengthening; and advice to perform exercise regularly. The therapist will treat the participants once a week for a 5-week period, each session will last 40 minutes. Besides the standard care, the therapist will perform cardia mobilization, pylori mobilization, Oddi's sphincter mobilization,duodenum-jejunum valve mobilization, ileocecal valve mobilization, global technique for the liver, global hemodynamic technique. Each technique will last 1 minutes, with the two last ones repeated 10 times.The placebo intervention involves light touch at the same regions of the techniques as above, and no intention on the part of the therapist to impart any therapeutic technique.
Who Masked: Outcomes Assessor
Masking Description: The evaluator will be blind as he will not be present during the intervention. As well as the care provider will not be present during the assessor activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The participants will receive standard care physiotherapy plus active visceral manipulation
  Interventions: Other: Active Visceral Manipulation; Other: Standard care physiotherapy
- Control Group (Placebo Comparator): The participants will receive standard care physiotherapy plus placebo visceral manipulation
  Interventions: Other: Standard care physiotherapy; Other: Placebo Visceral Manipulation

INTERVENTIONS:
Other: Active Visceral Manipulation — Visceral manipulation techniques consists of deep manual pressure in certain points of the abdomen and the amount of pressure will be respected according to the participant discomfort or pain. It will be performed cardia mobilization, pylori mobilization, Oddi's sphincter mobilization, duodenum-jejunum valve mobilization, ileocecal valve mobilization, global technique for the liver, global hemodynamic technique. Each technique will last 1 minutes, with the two last ones repeated 10 times.
  Other Names: Active Visceral Mobilization; Direct Visceral Mobilization
  Arms: Experimental Group
Other: Standard care physiotherapy — The care includes advice for correct postures to perform daily activities; abdominal, pelvic and lumbar muscles re-training and strengthening; and advice to perform at least 20 minutes' walk three times a week. The therapist will treat the participants once a week for a 5-week period. All treatment session will last 40 minutes.
  Other Names: Conventional physiotherapy
Other: Placebo Visceral Manipulation — The placebo intervention involves light touch at the same regions of the techniques the active visceral manipulation, and no intention on the part of the therapist to impart any therapeutic technique
  Other Names: Placebo Visceral Mobilization; Indirect Visceral Mobilization
  Arms: Control Group

SUMMARY:
Non-specific chronic low back pain is a common multifactorial condition common to the world population. It is defined as a pain and discomfort located below the ribs and above the gluteal folds that may or may not have referred pain in the leg for more than 12 weeks. Visceral manipulation is a manual therapy technique that aims to normalize mechanical, vascular and neurological dysfunctions of the viscera with the objective of improving its functioning. Visceral dysfunction may potentially activate or exacerbate the symptoms of low back pain in the presence of compromised movements between the internal organs and its connective tissues. There are two ways in which a change in visceral mobility could interfere with low back pain, referred visceral pain and central hypersensitivity. The first occurs due to neural convergence, since there is no spinocortical tract that only sends visceral or somatic afferences, its afferences are crossed in the dorsal horn of the spinal cord. The second is that the prolonged and continuous activation of nociceptors, due to the alteration in the mobility of the gastrointestinal and urinary system, can generate central hypersensitivity. Therefore, the investigators hypothesized that through the visceral manipulation the fascial adherences would lyse and the visceral spasms would demise, reducing the peripheral input, thus, lessening pain in the low back.

DETAILED DESCRIPTION:
Ethical aspects: All volunteers will be informed about the experimental procedures that will be submitted, as well as the fact that these do not affect the participant's health. The participants will also be clarified as to the secrecy of the information collected during the study performance, protecting the identities of the participants. After agreeing to participate in the research, each volunteer will sign the Informed Consent Term, according to resolution 196/96 and update in resolution 466 in 2012 of the National Health Council.

Risks:The interventions offer no harm to the participant's health. There is the possibility of the participant feeling pain and / or tickling during abdominal palpation. If these sensations occur, the procedure will be stopped and tried again. If sensations persist and the participant can not support them the session will be rescheduled or the participant will be disconnected from the study as there is no other way to carry out the proposed therapy.

Benefits:There may be no direct or immediate benefits, however, it is expected that the proposed treatment will improve lumbar pain.

This study does not offer any type of health insurance, and also, it is the responsibility of the participant to get around and bear the costs of transportation to the place of collection of data.

Confidentiality and privacy of research participants will be guaranteed during all phases of the research. At any time the participant can withdraw consent to participate in the research without any kind of penalty.

The research team is committed to making the search results public, whether favorable or not.

It is worth noting that the placebo intervention procedures will always be performed in association with an active treatment, which makes its use of less impact to the patient. In addition, all patients will be informed of the use of this procedure prior to the initiation of the survey.

Criteria for suspending research: This research will be suspended in the event of researchers' deaths, closure of the research site or termination of the Term of Science of the Partner Condition and / or no volunteer to participate in the research.

Financing This study will be funded by the researchers themselves.

Source of Patients: Patients with chronic low back pain will be referred for screening from online surveys, third party indications, and from patients on the waiting list of the Heath Center of the University of Sorocaba. The screening, assessment and evaluation will be performed at the Health Nucleus and in the Integrated Human Movement Laboratory of the University of Sorocaba.

Procedure: The researchers will inform the study objectives and procedures to all patients. If the participants agree to participate, the participants will sign an informed consent form. After that, a therapist will assess them for demographic data and baseline measures, such as pain level (0-10 Numerical Pain Rating Scale), disability associated with low back pain (Roland-Morris Disability Questionnaire), and function (0-10 Patient-Specific Functional Scale)

Random Allocation: One of the researchers will create a randomization code with 1:1 allocation radio using Excel for Windows software. The codes will be the words "E" for experimental or "P" for placebo, then ithe codes will be sealed on opaque envelopes, thus ensuring the concealed allocation of participants to groups. At the first encounter with the treating therapist, patients will choose one of the envelopes on a table and give it to the therapist. The therapist will open it in a different room from the patient and allocate the patient to the group according to the randomization schedule.

Interventions: The volunteers will be allocated in the Experimental group or the Control Group. In the Experimental, the participants will receive the Standard care physiotherapy plus Active visceral manipulation, while the Control will receive Standard care physiotherapy and Placebo visceral manipulation. The standard care physiotherapy lasts 40 minutes and the visceral mobilisation takes around 10 minutes.

Blinding: The assessor and the therapist will be blind to each others work. Therefore the assessor will not have knowledge of the treatment allocation and will perform three assessments, the pre assessment, immediately after the last treatment and 1 week after the treatment. Similarly, the therapist will not know the pre- and post-assessment intervention. In addition, there will be only one assessor and one therapist for the research to decrease bias. To test the blinding, after the last treatment session, the assessor will write on the patient's assessment chart which type of intervention (active or placebo) he thought the participant had received. These codes will be later compared with the randomization codes.

Statistical methods: Statistical analysis will be used SPSS (Statistical Package for Social Sciences) v.19.0. Initially the Kolmogorov-Smirnov test will be performed. If the data are normal, parametric tests will be applied, if the distribution is non-normal, non-parametric tests will be used. It will be calculated from the effect size, by means of the difference between the means of the pre-intervention evaluation and the post-intervention evaluation. In all analyzes, a critical level of 5% (p <0.05) will be set.

ELIGIBILITY:
Inclusion Criteria:

* primary complaint of chronic non-specific low back pain (more than 12 weeks);
* pain symptoms in the low back with a score ≥ 2/10 on the 0-10 Numerical Pain Rating Scale (12);
* aged 18-80;
* history of surgery in the abdominopelvic region for more than 6 months;
* history of visceral dysfunction (e.g., constipation and reflux); and
* no known or suspected serious spinal pathology (e.g., metastasis, inflammatory or infective diseases of the spine, causa equine syndrome, canal stenosis, spinal fracture).

Exclusion Criteria:

* no nerve root compromise evidenced by at least two of the following: (1) myotomal weakness, (2) dermatomal or widespread sensory loss, (3) hyporeflexia or hyperreflexia of the lower limb reflexes;
* no spinal surgery within the preceding 6 months;
* no vascular abnormality such as abdominal aortic aneurysms;
* not currently receiving chiropractic, osteopathic or other physical therapy;
* not pregnant or suspect being pregnant;
* not currently in an acute inflammatory phase of known gastrointestinal or urinary diseases (such as cholecystitis, renal calculi, peritonitis, appendicitis);
* not currently taking medications that significantly alter gut motility;
* not currently taking medications (such as oral corticosteroids) which are known to increase the risk of intestinal perforation);
* no known gastrointestinal disease that associates with a risk of intestinal perforation (e.g. Chron's disease, diverticular disease, peptic ulcer disease);
* not taking anti-platelet medications such as warfarin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas V Santos, Principal Investigator — University of Sorocaba
Locations (2):
- Brazil (2):
  - Integrated Laboratory of Human Movement, University of Sorocaba, Sorocaba, São Paulo
  - Health Center, University of Sorocaba, Sorocaba, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BARRAL, J.-P .; MERCIER, P. Visceral Manipulation. [Sl: sn].
- [Background] Bove GM, Chapelle SL. Visceral mobilization can lyse and prevent peritoneal adhesions in a rat model. J Bodyw Mov Ther. 2012 Jan;16(1):76-82. doi: 10.1016/j.jbmt.2011.02.004. Epub 2011 Apr 9. PMID 22196431
- [Background] Cervero F. Visceral pain-central sensitisation. Gut. 2000 Dec;47 Suppl 4(Suppl 4):iv56-7; discussion iv58. doi: 10.1136/gut.47.suppl_4.iv56. No abstract available. PMID 11076916
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Nascimento PR, Costa LO. Low back pain prevalence in Brazil: a systematic review. Cad Saude Publica. 2015 Jun;31(6):1141-56. doi: 10.1590/0102-311X00046114. Epub 2015 Jun 1. English, Portuguese. PMID 26200363
- [Background] Nusbaum L, Natour J, Ferraz MB, Goldenberg J. Translation, adaptation and validation of the Roland-Morris questionnaire--Brazil Roland-Morris. Braz J Med Biol Res. 2001 Feb;34(2):203-10. doi: 10.1590/s0100-879x2001000200007. PMID 11175495
- [Background] Panagopoulos J, Hancock MJ, Ferreira P, Hush J, Petocz P. Does the addition of visceral manipulation alter outcomes for patients with low back pain? A randomized placebo controlled trial. Eur J Pain. 2015 Aug;19(7):899-907. doi: 10.1002/ejp.614. Epub 2014 Nov 7. PMID 25378096
- [Background] REZENDE, RPDB; GABRIEL, A. Relationship between Clinic and Osteopathy. Rev. Soc. Bras. Clin. Avg, v. 6, n. 5, p. 194-196, 2008.
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533
- [Background] STRATFORD P, GILL C, WESTAWAY M, ET AL. A. DISABILITY AND CHANGE ON INDIVIDUAL PATIENTS: A REPORT OF A PATIENT SPECIFIC. . .Patient-Specific Functional Scale Patient-Specific Functional Scale. Physiother Can 1995; 47: 258-63. , V. 47: 258-63., P. 3, 1995.
- [Background] Tozzi P, Bongiorno D, Vitturini C. Low back pain and kidney mobility: local osteopathic fascial manipulation decreases pain perception and improves renal mobility. J Bodyw Mov Ther. 2012 Jul;16(3):381-391. doi: 10.1016/j.jbmt.2012.02.001. Epub 2012 Mar 3. PMID 22703751
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited through third party referral from the Health Center of the University of Queensland. The date of recruitment was from 06/01/2017 to 06/16/2017. The participants usually knew about the study through advertisement on online social media or through folders on the Health Center clinic.
Pre-assignment Details: There were no events that occur after participant enrollment, but prior to assignment of participants to a group
Groups:
- Experimental Group: 10 participants received standard care physiotherapy plus active visceral manipulation
  Active Visceral Manipulation: Visceral manipulation techniques consists of deep manual pressure in certain points of the abdomen and the amount of pressure will be respected according to the participant discomfort or pain. It will be performed cardia mobilization, pylori mobilization, Oddi's sphincter mobilization, duodeno-jejunal valve mobilization, ileocecal valve mobilization, global technique for the liver, global hemodynamic technique. Each technique will last 1 minutes, with the two last ones repeated 10 times.
  Standard care physiotherapy: The care includes advice for correct postures to perform daily activities; abdominal, pelvic and lumbar muscles re-training and strengthening; and advice to perform at least 20 minutes' walk three times a week. The therapist will treat the participants once a week for a 5-week period. All treatment session will last 40 minutes.
- Control Group: 10 participants received standard care physiotherapy plus placebo visceral manipulation
  Standard care physiotherapy: The care includes advice for correct postures to perform daily activities; abdominal, pelvic and lumbar muscles re-training and strengthening; and advice to perform at least 20 minutes' walk three times a week. The therapist will treat the participants once a week for a 5-week period. All treatment session will last 40 minutes.
  Placebo Visceral Manipulation: The placebo intervention involves light touch at the same regions of the techniques the active visceral manipulation, and no intention on the part of the therapist to impart any therapeutic technique
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 10 | 10
Completed | 9 | 7
Not Completed | 1 | 3
Not completed — Lack of time to participate | 1 | 0
Not completed — Ran over by a car | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: 20 participants with chronic low back pain and visceral dysfunction
Groups:
- Experimental Group: The participants received standard care physiotherapy plus active visceral manipulation
  Active Visceral Manipulation: Visceral manipulation techniques consists of deep manual pressure in certain points of the abdomen and the amount of pressure will be respected according to the participant discomfort or pain. It will be performed cardia mobilization, pylori mobilization, Oddi's sphincter mobilization, duodeno-jejunal valve mobilization, ileocecal valve mobilization, global technique for the liver, global hemodynamic technique. Each technique will last 1 minutes, with the two last ones repeated 10 times.
  Standard care physiotherapy: The care includes advice for correct postures to perform daily activities; abdominal, pelvic and lumbar muscles re-training and strengthening; and advice to perform at least 20 minutes' walk three times a week. The therapist will treat the participants once a week for a 5-week period. All treatment session will last 40 minutes.
- Control Group: The participants received standard care physiotherapy plus placebo visceral manipulation
  Standard care physiotherapy: The care includes advice for correct postures to perform daily activities; abdominal, pelvic and lumbar muscles re-training and strengthening; and advice to perform at least 20 minutes' walk three times a week. The therapist will treat the participants once a week for a 5-week period. All treatment session will last 40 minutes.
  Placebo Visceral Manipulation: The placebo intervention involves light touch at the same regions of the techniques the active visceral manipulation, and no intention on the part of the therapist to impart any therapeutic technique
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.39) | 40.5 (12.12) | 40.5 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 10 | 10 | 20
Visceral dysfunction [Count of Participants; unit: Participants] — Visceral dysfunction is considered to be symptoms of constipation or any kind of surgery that the participant had undergone through.
  Participants | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain After 6 Weeks of Intervention
Description: An 11-point Numeric Pain Rating Scale (NPRS) will be used, where 0 is equivalent to "no pain" and 10 to "unbearable pain"
Time Frame: 6 weeks
Population: 20 participants with low back pain and visceral dysfunction
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 10 | 10
units on a scale
  pre-intervention | 6.50 (2.33) | 6.00 (0.92)
  post-intervention | 1.50 (2.42) | 3.50 (2.94)
  1 week follow-up | 1.80 (2.93) | 3.30 (3.20)

2. Secondary Outcome: Low Back Mobility Using the Schober Test After 6 Weeks of Intervention
Description: The Schober test consists of extending a tape measure on the spinal column, between the two posterior superior iliac spines and up to 10 cm above this, with the individual in a neutral position. Then, the patient is asked to do anterior flexion of the trunk, then the therapist will measure the distance of the marked points, in patients without changes of mobility should increase at least 5 cm. Increases smaller than 5 cm indicate that the test is positive, decreased mobility of the lumbar spine.
Time Frame: 6 weeks
Population: 20 participants with chronic low back pain and visceral dysfunction
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 10 | 10
centimeters
  pre-intervention | 14.75 (0.78) | 15.31 (1.00)
  post-intervention | 15.88 (1.09) | 15.30 (0.63)
  1 week follow-up | 15.71 (1.04) | 15.11 (1.04)

3. Secondary Outcome: Disability Due to Low Back Pain After 6 Weeks of Intervention
Description: The Roland Morris Disability Questionnaire consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/activity, sleep/rest, psychosocial, household management, eating and pain frequency. It is designed to take approximately 5 minutes to complete, without any assistance from the administrator.
  The respondent is presented with each statement and asked if they feel the statement is descriptive of their own circumstance on that day. For example, the first statement is 'I stay at home most of the day because of the pain in my back'. If the respondent feels that this statement applies to them they 'tick' the statement, otherwise they leave it blank. To score the responses, a practitioner need only add up the number of items ticked. There is no weighting applied to the statements, therefore the score can range from 0 (no disability) to 24 (maximal disability).
Time Frame: 6 weeks
Population: 20 participants with chronic low back pain and visceral dysfunction
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 10 | 10
points
  pre-intervention | 12.00 (4.15) | 9.20 (6.16)
  post-interverntion | 6.60 (6.12) | 5.10 (4.48)
  1 week follow-up | 5.30 (5.06) | 3.80 (4.53)

4. Secondary Outcome: Functional Activity After 6 Weeks of Intervention
Description: he Patient-Specific Functional Scale (PSFS) is a self-reported, patient-specific outcome measure, designed to assess functional change, primarily in patients presenting with musculoskeletal disorders Patients are asked to identify up to five important activities they are unable to perform or are having difficulty with as a result of their problem i.e. putting socks on. In addition to identifying the activities, patients are asked to rate, on an 11-point scale, the current level of difficulty associated with each activity. Following the intervention, patients are asked again to rate the activities previously identified and are given the chance to nominate new problematic activities that might have arisen during that time."0" represents "unable to perform". "10" represents "able to perform at prior level".
  Patients select a value that best describes their current level of ability on each activity assessed. Lower scores mean a worse outcome, higher scores mean a better outcome.
Time Frame: 6 weeks
Population: 20 participants with chronic low back pain and visceral dysfunction
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 10 | 10
units on a scale
  pre-intervention | 5.90 (3.05) | 4.10 (3.08)
  post-intervention | 3.20 (2.71) | 4.50 (3.29)
  1 week follow-up | 3.90 (3.33) | 3.90 (2.77)

ADVERSE EVENTS:
Time Frame: The adverse effects were collected before and after each session. A total of 5 weeks.
Description: The patients were asked by the treating physiotherapist about adverse effects such as sore muscles, back pain and abdominal discomfort. The therapist took note on a blank paper corresponding to the participant identification number.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=10) | Control Group (N=10)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle soreness (Musculoskeletal and connective tissue disorders) | 10 | 10
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
High dropout rate for the control group compromised statistical power; Unreliability of the placebo technique.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03101020/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03101020/SAP_001.pdf